CLINICAL TRIAL: NCT07090889
Title: A Combined Single and Multiple Ascending Dose Phase 1a/1b, Double-blind, Placebo-Controlled, and Food-effect Study to Evaluate the Safety and Pharmacokinetics of Oral KM-023 in Healthy Participants. Followed by a 3-month Open Label Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Oral KM-023 in Olmsted Syndrome Patients
Brief Title: Study of KM-023 in Healthy Volunteers and Patients With Olmsted Syndrome.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kamari Pharma Ltd (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KM-023-101
Record Dates: First submitted 2025-05-08; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Olmsted Syndrome
MeSH Terms: interventions — 3-(3-ethyl-5-isopropyl-2,6-dioxo-1,2,3,6-tetrahydropyrimidine-4-carbonyl)-5-methylbenzonitrile

STUDY DESIGN:
Intervention Model Description: The study includes two parts:
  Part A- a Single Ascending Dose (SAD) part followed by a Multiple Ascending Dose (MAD) part, Placebo- controlled Part B- Open Label
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A SAD (Single Ascending Dose) (Active Comparator): Up to 4 cohorts of 8 healthy participants
  Interventions: Drug: KM-023; Drug: Placebo
- Part A MAD (Multiple Ascending Dose) (Active Comparator): 3 cohorts of 8 healthy participants.
  Interventions: Drug: KM-023; Drug: Placebo
- Part B- OS patients (Active Comparator): up to 8 participants with OS, receiving KM-023 for 12 weeks.
  Interventions: Drug: KM-023

INTERVENTIONS:
Drug: KM-023 — solution for oral administration
Drug: Placebo — solution for oral administration
  Arms: Part A MAD (Multiple Ascending Dose); Part A SAD (Single Ascending Dose)

SUMMARY:
The trial is conducted in order to assess the safety of KM-023 and to observe what effects, both beneficial and adverse, it has on the body, and the way the body absorbs and eliminates KM-023, first in healthy participants, then in Olmsted Syndrome patients. In addition, the study will examine the presence of KM-023 in the different layers of the skin. Finally, the efficacy of KM-023 will be investigated in Olmsted Syndrome patients.

The first part of this trial will be conducted with healthy participants in France, then after its completion, the second part of the trial will be conducted with Olmsted Syndrome patients in France and the United Kingdom.

The first part of the trial is itself divided in two parts: first, a series of single doses will be given to groups of healthy participants, then other groups of healthy participants will be given repeated doses of KM-023 twice daily for 5 days.

The participants will be hospitalized approximately 2 days for the investigation of single doses, and approximately 8 days for the investigation of the multiple doses.

Some participants will receive the KM-023, and other will receive a placebo, which is a non-active product.

Four (4) different dose levels will be given in the trial part studying single administration, and 3 different dose levels in the trial part studying repeated administrations. The trial will start with the lowest doses, and the dose levels will be gradually increased after the safety and tolerability of the previous dose level has been assessed by a group of experts (including physicians). In order to assess the safety, a series of examinations will be conducted, including taking blood samples. Blood samples will also be collected a regular timepoints in order to evaluate the changes in concentration of KM-023 in blood over time. One group of participants will receive a single dose of KM-023 twice: once after fasting, and once with a meal, to check any effect of food on the concentration of KM-023 in blood.

In the second part of the trial, Olmsted Syndrome patients will take KM-023 twice daily, for a duration of 12 weeks.

There will be a first hospitalization day, during which the patients will receive the study drug, and will be taught how to self-administer KM-023 at home during the ambulatory periods. Safety and efficacy tests will be performed, and the concentration of KM-023 in blood will be monitored. Patients will then go back home with their treatment, to be taken every day. After the first hospitalization day, there will be five visits (two of them will be 1-day hospitalization periods), to monitor the safety and tolerability, the efficacy, and the concentration of KM-023 in blood. Between the hospitalization visits, the clinical teams will call the patients at home on a regular basis to check the safety and tolerability.

The duration of participation, including the selection period and the follow-up period, is a maximum 36 days when only one dose is given, 51 days when the dose is given on two occasions to assess the effect of food, 40 days when treatment is given twice daily for 5 days, and 18 weeks in the case of Olmsted Syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Healthy female and male participants.
* Female participants of non-childbearing potential, childbearing potential and males capable of fathering a child must meet the contraception requirements.
* Non-smoking and no use of any tobacco or nicotine products (by declaration) for a period of at least 1 month prior to screening visit.
* Not using prescription medication 14 days prior to admission; and 7 days prior to admission for over the counter (OTC) medication/vitamins/supplements.
* Must not be taking any medication that could potentially impair hepatic or renal function at the time of screening.
* No history of alcohol or other drugs of abuse.
* Body Mass Index (BMI) of 18.0 to 32.0 kg/m2 (inclusive); and a total body weight >50.0 kg (110 lbs) and <100.0 kg (220 lbs) at screening and Day -1.
* No vaccines given within 14 days of dosing.
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.

Part B

* Read, understood, and signed an ICF before any investigational procedure(s) are performed.
* Clinical diagnosis of OS, with confirmed TRPV3 or PERP mutation, and visible palmoplantar keratoderma.
* Stable medical condition over the previous 1 month.
* Willingness and ability to comply with the treatment and follow-up visits.
* Willingness to refrain from current treatments, in compliance with the list of prohibited medications.
* No contraindications to study medication as determined by the Investigator.
* Female participants of non-childbearing potential, childbearing potential and males capable of fathering a child must meet the contraception requirements.
* Negative serum pregnancy test at screening, and negative urinary pregnancy test at Day -1.

Exclusion Criteria:

Part A

* Participants who are staff members at the investigational site directly involved in conducting the study.
* Evidence or history of clinically relevant hepatic, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males within 6 months of screening.
* Screening supine BP ≥145 mm Hg (systolic) or ≥90 mm Hg (diastolic)
* Participants with any abnormalities in clinical laboratory tests, and serology results, at screening, considered by the study physician as clinically significant.
* Pregnant or breastfeeding female participants.
* Participants who donated blood or received blood or plasma derivatives in the 30 days preceding study drug administration.
* Dosed in another clinical trial within at least 10 tissue half-lives prior to dosing or 4 months.
* Known relevant allergy to any drug or excipients in the formulation
* Participants with any acute medical situation (e.g., acute infection) within 48h of screening or start of dosing, which is considered of significance by the Investigator.
* Major surgery within the last 3 months or any planned surgery during the trial.
* Unwilling or unable to comply with all scheduled visits, treatment plan, laboratory tests and other study procedures and the restrictions described in the protocol.
* Any other condition or previous therapy that, in the opinion of the Investigator or their designee, would render the participant unsuitable for this study, including an inability to fully comply with the study protocol requirements or a likelihood of noncompliance with study procedures.

Part B

* The presence of other significant dermatological conditions that could interfere with the evaluation of the study treatment's safety and efficacy.
* Active or uncontrolled infections (e.g., sepsis, tuberculosis, hepatitis B or hepatitis C at the screening visit, human immunodeficiency virus[HIV]) that could complicate participation in the study.
* Any medical or active psychological condition or any clinically relevant laboratory abnormalities, such as, but not limited, to elevated ALT or AST (> 3 × ULN) in combination with elevated bilirubin (> 2 × ULN), at the screening/baseline visit.
* Diabetic foot ulcers.
* Patient is unwilling to refrain from using prohibited medications during the clinical trial.
* Currently participating or participated in any other clinical trial of an IMP or device, within the past 4 months before the screening visit.
* Cutaneous infection or another underlying condition of the skin which may impact the assessments or trial participants.
* Cutaneous infection of the area to be treated with IMP within 2 weeks before the screening visit or any infection of treatment area requiring treatment with oral, parenteral antibiotics, antivirals, antiparasitics or antifungals or any topical within 2 weeks before the screening visit.
* Pregnant or breastfeeding patient.
* Having received any of the prohibited treatments in Table 2 within the specified timeframe before inclusion.
* Known relevant allergy to any drug or excipients in the formulation.
* Major surgery within the last 3 months, or minor surgery (requiring local anesthetic) during last 1 month, or any planned surgery during the trial.
* Unwilling or unable to comply with all scheduled visits, treatment plan, laboratory tests and other study procedures and the restrictions described in the protocol.
* Any other condition or previous therapy that, in the opinion of the Investigator or their designee, would render the patient unsuitable for this study, including an inability to fully comply with the study protocol requirements or a likelihood of noncompliance with study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and other safety-related events. | Part A- SAD(Single Ascending Dose) day 8, MAD (Multiple Ascending Dose) day 12 Part B- Day 112.

SECONDARY OUTCOMES:
Reduction in target plantar callus thickness from baseline to visit at Week 12. (Part B only) | 12 weeks
Reduction in target plantar callus size from baseline to visit at Week 12. (Part B only) | 12 weeks
Clearance of the lesions, assessed by change from baseline to W4, 8 and 12 in Investigator Global Assessment (IGA) score. (Part B only) | 12 weeks
Peak Plasma Concentration (Cmax) | Part A - SAD (Single Ascending Dose) Day 8; MAD (Multiple Ascending Dose) Day 12; Part B - Day 112.
  Peak plasma concentration (Cmax) of the study drug.
Time to Reach Peak Plasma Concentration (Tmax) | Part A - SAD Day 8; MAD Day 12; Part B - Day 112.
  Time to reach maximum observed plasma concentration (Tmax) of the study drug.
Area Under the Plasma Concentration-Time Curve (AUC) | Part A - SAD Day 8; MAD Day 12; Part B - Day 112.
  Area under the plasma concentration-time curve (AUC) of the study drug.
Dose Proportionality of Pharmacokinetic Parameters | Part A - SAD Day 8; MAD Day 12; Part B - Day 112.
  Dose proportionality assessment of pharmacokinetic parameters (Cmax and AUC) within the administered dose range.

OTHER OUTCOMES:
Quantitative analysis of KM-023 distribution across skin layers at various timepoints, utilizing imaging mass spectrometry with matrix-assisted laser desorption/ionization (MALDI). | Part A- SAD(Single Ascending Dose) day 8, MAD (Multiple Ascending Dose) day 12 Part B- Day 112.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial, Rennes, France